CLINICAL TRIAL: NCT00679575
Title: Statins and Risk of Myocardial Infarction in Real Life in France
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Russel Esterline, AstraZeneca
Other Study IDs: NIS-CFR-CRE-2007/1
Record Dates: First submitted 2008-05-15; First posted 2008-05-19 (Estimated); Last update posted 2010-12-08 (Estimated); Status verified 2010-12

CONDITIONS: Myocardial Infarction
Keywords: statins; myocardial infarction; case-referent study; France
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Cases : Patients with a first myocardial infarction
- 2: Referents : Patients recruited by a GP during a routine consultation

SUMMARY:
The main objective of this case-referent study is to assess the impact of statins usage on the risk of having a first myocardial infarction (MI) in a real life situation in France

ELIGIBILITY:
Inclusion Criteria:

* Patients can speak French or English
* Patients can be interviewed by telephone
* Place of usual residence in the area of recruitment

Exclusion Criteria:

* Patients refusing to participate in the study
* Patients who cannot be reached by telephone
* Previous history of myocardial infarction

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cases : Patients recruited by a cardiologist in hospital / Referents : Patients recruited by a GP, community sample
Sampling Method: Probability Sample
Enrollment: 13171 (Actual)
Dates: Start 2007-03; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Assess the impact of the different statins (molecules) usage on the risk of having a first myocardial infarction in a real life situation in France | in 2011

SECONDARY OUTCOMES:
Assess the interaction between statin treatment and risk factors such as cholesterol, age, gender, tobacco, alcohol, co-prescriptions, co-morbidities | in 2011
Assess the populational impact of statins usage on the risk of having a first myocardial infarction | in 2011
Assess the risk of having a first myocardial infarction according to high and low dosages of statins | in 2011

CONTACTS AND LOCATIONS:
Overall Officials: Lucien Abenhaim, Study Chair — LA-SER29, rue du Faubourg Saint-Jacques75014 Paris
Locations (56):
- France (56):
  - Research Site, Ambilly
  - Research Site, Angers
  - Research Site, Arles
  - Research Site, Bagnols-sur-Cèze
  - Research Site, Bayonne
  - Research Site, Béziers
  - Research Site, Boulogne-sur-Mer
  - Research Site, Bourgoin
  - Research Site, Bron
  - Research Site, Cambo-les-Bains
  - Research Site, Cenon
  - Research Site, Châteauroux
  - Research Site, Clermont-Ferrand
  - Research Site, Colmar
  - Research Site, Crest
  - Research Site, Dijon
  - Research Site, Draguignan
  - Research Site, Eaubonne
  - Research Site, Firminy
  - Research Site, Forbach
  - Research Site, Fréjus
  - Research Site, Gleizé
  - Research Site, Grasse
  - Research Site, Guéret
  - Research Site, La Rochelle
  - Research Site, Langres
  - Research Site, Laon
  - Research Site, Le Coudray
  - Research Site, Le Mans
  - Research Site, Le Puy-en-Velay
  - Research Site, Mayenne
  - Research Site, Millau
  - Research Site, Montélimar
  - Research Site, Montfermeil
  - Research Site, Montpellier
  - Research Site, Nîmes
  - Research Site, Orange
  - Research Site, Orléans
  - Research Site, Paris
  - Research Site, Pau
  - Research Site, Perpignan
  - Research Site, Puilboreau
  - Research Site, Rueil-Malmaison
  - Research Site, Rumilly
  - Research Site, Saint Amand Monrond
  - Research Site, Saint Jean Des Verges
  - Research Site, Saint-Estève
  - Research Site, Sallanches
  - Research Site, Salon-de-Provence
  - Research Site, Sens
  - Research Site, Thonon-les-Bains
  - Research Site, Toulouse
  - Research Site, Tours
  - Research Site, Tulles
  - Research Site, Valence
  - Research Site, Villefranche-de-Rouergue